Study Title: Ketamine for Suicidality in Bipolar Depression

NCT number: NCT01944293

Date: 5/14/2019

## Statistical methods

The intent-to-treat analysis included all randomized participants. We used R software (r-project.org) and SPSS version 23 (IBM, Armonk, NY, USA). Univariate tests compared groups on baseline characteristics. Histograms were inspected for normality. The primary hypothesis was tested using a linear regression model of day 1 SSI (SSIday1) with baseline SSI (SSIBL) and treatment as the predictors: SSIday1 ~ SSIBL + treatment. Secondary analyses tested treatment effect on response and remission. Effect size calculations used Cohen's d and number needed to treat (NNT). We used regression models analogous to that for SSI to test effects on depression, mania, and anxiety. The POMS was analyzed with a generalized least squares (GLS) model over its three assessment time-points. Since at randomization only one subject was not taking psychiatric medications and only one subject had baseline SSI <8, we did not adjust for the randomization strata. We tested a repeated measures analysis of covariance (ANCOVA) model of SSI, including 230 minute and day 1 assessments, analyzed response to the openlabel ketamine infusion, and tested the correlation between change in depressive symptoms and change in SSI. We plotted mean SSI during the 6-week follow-up in those randomized to ketamine and performed paired t tests of the score each week compared to baseline. We investigated infusion effects on neurocognition and explored relationships of clinical variables with CAR, serum BDNF, and postinfusion plasma ketamine, norketamine and dehydronorketamine.31 Safety analyses investigated dissociative, psychotomimetic and cardio-respiratory effects.